CLINICAL TRIAL: NCT01748955
Title: SSRI Versus Bupropion in High-Risk Major Depressive Disorder
Brief Title: Paroxetine/Bupropion in Depression With Suicide Attempt or Thoughts: fMRI Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5933R; K23MH076049 (NIH)
Record Dates: First submitted 2012-09-20; First posted 2012-12-13 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Depression; Suicidal Ideation
Keywords: Major Depressive Disorder; MDD; Reward; BOLD signal; Suicide
MeSH Terms: conditions — Depression; Suicidal Ideation; Depressive Disorder, Major; Suicide | interventions — Paroxetine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupropion (Active Comparator): Participants will receive bupropion XL for 8 weeks.
  Interventions: Drug: Bupropion XL for Major Depressive Episode
- paroxetine CR (Active Comparator): Participants will receive Paroxetine CR for 8 weeks.
  Interventions: Drug: Paroxetine CR for Major Depressive Episode

INTERVENTIONS:
Drug: Paroxetine CR for Major Depressive Episode — Dosage will be 25mg every day for 2 weeks, then 37.5mg every day for 2 weeks, and then optional increase to 50mg every day for the remainder of treatment.
  Other Names: Paxil CR
  Arms: paroxetine CR
Drug: Bupropion XL for Major Depressive Episode — Dosage will be 150mg every day for 2 weeks, then 300mg every day for 2 weeks, and then optional increase to 450mg every day for the remainder of treatment.
  Other Names: Wellbutrin XL
  Arms: Bupropion

SUMMARY:
This study uses functional magnetic resonance imaging (fMRI) to investigate the effects of two different antidepressant medications (Paxil CR versus Wellbutrin XL) on reward processing in depressed patients who have attempted suicide or are currently experiencing suicidal thoughts.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common and serious psychiatric illness. It is among the leading causes of disability and is the psychiatric disorder most often associated with suicide. The treatment of MDD with antidepressant medication remains largely trial and error. Little empirical evidence exists to guide the treatment of MDD when suicide risk is a major factor.

The study uses functional magnetic resonance imaging (fMRI) to compare the effects of paroxetine, an SSRI, versus bupropion, a non-SSRI, on brain activity in depressed patients with a past suicide attempt and/or current suicidal thoughts. Participants are randomly assigned to either paroxetine or bupropion treatment for 8 weeks, with fMRI scans involving a reward processing task at baseline and Week 8. Weekly study visits include interviews with a psychologist, self-report scales, and medication monitoring. All participants will then be offered 4 additional months of open clinical treatment. If original medication assignments prove to be ineffective, participants will have the option to switch to another medication. After completing the study, participants will be referred for ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient suffering from an episode of major depressive disorder (MDD)
2. Age range 18-65 years
3. History of a past suicide attempt or score > 2 on HDRS item #3 (suicide) at in-person screening interview. Patients with suicidal plan or intent will only be enrolled as inpatients if independent inpatient treatment team agrees with the plan to enroll the patient.
4. Patients 60 years of age and older must score at least 25 on MMSE at screening.
5. Patients 60 years of age and older must have a normal ECG within the past year.

Exclusion Criteria:

1. Bipolar disorder; current psychotic symptoms; bulimia or anorexia that is current or within the past year, or current purging at least twice a week for three months; persons already taking SSRIs or bupropion for other indications (such as anxiety disorders).
2. Primary disorder is an anxiety disorder such as Panic disorder/GAD/OCD/ Social anxiety disorder, with secondary depression.
3. Drug or alcohol dependence within past six months; persons with current drug or alcohol abuse may be enrolled if this is assessed as being of lesser importance than the major depressive episode.
4. Blood pressure reading ≥ 140/90
5. Active and/or unstable medical problems including a significant risk for seizures
6. Antipsychotic medication required
7. Patients who have become hypomanic or manic on antidepressants
8. Contraindication to the use of an SSRI or bupropion, or currently using Zyban. Anorexia nervosa in remission at least one year is not an exclusion.
9. Failure to respond to adequate trials of 3 SSRIs or paroxetine or bupropion in the last 2 years (failure to respond to therapeutic trial defined as: at least 2/3 maximal PDR dose for at least 6 weeks).
10. Lacks capacity to consent
11. Pregnancy, lactation, or plans to conceive during the course of study participation.
12. Patients currently on effective treatment, who require adjunctive antipsychotic or mood stabilizing medication, or who are unlikely to respond to single agent treatment for depression will be excluded.
13. Patients with ferrous metal implants in their bodies, or a history of claustrophobia that precludes MRI, will be excluded.
14. Patients assessed as being unlikely to tolerate the maximum 2-week delay to start of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Grunebaum, M.D., Principal Investigator — Columbia University/NY State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Grunebaum MF, Ellis SP, Duan N, Burke AK, Oquendo MA, John Mann J. Pilot randomized clinical trial of an SSRI vs bupropion: effects on suicidal behavior, ideation, and mood in major depression. Neuropsychopharmacology. 2012 Feb;37(3):697-706. doi: 10.1038/npp.2011.247. Epub 2011 Oct 12. PMID 21993207
- See also: Click here for the Columbia University Psychiatry Clinical Trials Web site — http://columbiapsychiatry.org/clinical-trials
- See also: MIND Clinic for Mood and Personality Disorders — http://www.columbiapsychiatry.org/mind/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion | Paroxetine CR
Started | 6 | 9
Completed | 3 | 4
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Paroxetine CR | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Contrast of Parameter Estimates (COPE)
Description: % change in COPE = (Post-treatment COPE - Pre-treatment COPE) / Pre-treatment COPE COPE is measured during Monetary Incentive Delay Task.
  Task conditions are:
  Reward= BOLD signal when subject wins 5 cents vs. wins 0 cents Punishment= BOLD signal when subject loses 5cents vs. loses 0 cents
Time Frame: Measured at Baseline (pre-treatment) and Week 8 (post-treatment)
Population: Major depressive disorder with suicidal thoughts or past suicide attempt.
Measure: Mean (Full Range); unit: Percentage change
Arm/Group | Bupropion | Paroxetine CR
Number analyzed (Participants) | 3 | 4
Percentage change
  ACC Reward | 0.29 [-1.74 to 2.90] | -2.12 [-7.38 to 0.46]
  ACC Punishment | -1.19 [-2.15 to -0.30] | -1.33 [-2.49 to -0.86]
  Amygdala Reward | -0.90 [-2.38 to 0.18] | -0.87 [-1.27 to -0.65]
  Amygdala Punishment | -0.32 [-1.53 to 0.93] | -0.66 [-1.22 to -0.13]

2. Secondary Outcome: Change in Suicidal Ideation (SSI Score)
Description: Beck Scale of Suicidal Ideation Minimum Value = 0 Maximum Value = 38 Higher score is more severe suicidal thoughts
Time Frame: Measured at Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion | Paroxetine CR
Number analyzed (Participants) | 3 | 4
units on a scale
  Baseline | 11 (4.4) | 4.8 (3.5)
  Week 8 | 3.3 (3.1) | 0.3 (0.5)

ADVERSE EVENTS:
Time Frame: 4 years, 0 months.
Arm/Group | Bupropion | Paroxetine CR
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No